CLINICAL TRIAL: NCT04356846
Title: A Phase I Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Preliminary Efficacy of the Oral BCL-2 Inhibitor LP-108 in Patients With Relapsed or Refractory B-cell Lymphoma
Brief Title: A Phase I Study of LP-108 in Patients With Relapsed or Refractory B-cell Lymphoma
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: The First Affiliated Hospital with Nanjing Medical University (Other)
Collaborators: Guangzhou Lupeng Pharmaceutical Company LTD. (Industry); Newave Pharmaceutical Inc (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LP-108-I-01
Record Dates: First submitted 2020-04-10; First posted 2020-04-22 (Actual); Last update posted 2023-05-01 (Actual); Status verified 2023-04

CONDITIONS: Non-Hodgkin Lymphoma; Chronic Lymphocytic Leukemia
MeSH Terms: conditions — Lymphoma, Non-Hodgkin; Leukemia, Lymphocytic, Chronic, B-Cell

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- R/R CLL (Experimental): Relapsed or Refractory Chronic Lymphocytic Leukemia Patients
  Interventions: Drug: LP-108 tablet
- R/R NHL (Experimental): Relapsed or Refractory B-cell Non-Hodgkin Lymphoma Patients, including SLL, FL, MZL, MCL, DLBCL, WM.
  Interventions: Drug: LP-108 tablet

INTERVENTIONS:
Drug: LP-108 tablet — Taken orally within 30 minutes after a meal at the designated dose, once daily.

SUMMARY:
This study is a multi-center, open-label, single-arm phase I clinical study of LP-108. Patients with relapsed or refractory chronic lymphocytic leukemia (CLL, arm A) and other B cell non-Hodgkin's lymphoma (NHL, Arm B). Each arm has a dose escalation phase (phase Ia) and expansion phase (phase Ib). During the dose escalation phase, the primary objectives are to define dose-limiting toxicity (DLT), maximum tolerated dose (MTD), and to explore a recommended phase II dose. Dose escalation is based on the classic "3 + 3" design, while accelerated titration is applied to the initial lower doses. After the RP2Ds are determined, additional patients will be enrolled in the expansion phase to further evaluation the safety, PK and preliminary efficacy of LP-108, each therapy can enroll 12-20 subjects.

ELIGIBILITY:
Inclusion Criteria:

* Per 2017 revised WHO lymphoma classification criteria, subject must have either:

  * (Arm A) Diagnosed with relapsed or refractory CLL and require treatment in the opinion of the Investigator.
  * (Arm B) Diagnosed with relapsed or refractory non-Hodgkin's lymphoma associated with B-cell proliferation (such as SLL \ MCL \ FL \ MZL \ DLBCL \ WM, etc.) in need of treatment.
* Subject has an Eastern Cooperative Oncology Group (ECOG) performance score less than or equal to 1.
* Subject must have adequate bone marrow function independent of growth factor support per local laboratory reference range at Screening.
* Subject must have adequate coagulation, renal, and hepatic function, per local laboratory reference range at Screening.
* All acute toxicity from previous anti-tumor treatment or surgery has been alleviated to NCI CTCAE 5.0 ≤ Grade 1.
* All enrolled patients should take medically approved contraceptives during the entire treatment period and within 90 days after the end of treatment.
* Subjects must be willing to provide valid diagnostic evidence or accept bone marrow biopsy before treatment and accept bone marrow biopsy after treatment start.
* Patients with NHL who have undergone autologous stem cell transplantation must complete the transplantation operation for more than 6 months when enrolled, and have sufficient bone marrow function without relying on growth factor stimulation.
* Volunteer and sign informed consent, willing to follow trial protocol.

Exclusion Criteria:

* According to the 2017 revised WHO Lymphoma Classification Criteria, patients diagnosed with the following diseases: Burkitt lymphoma or Burkitt-like lymphoma, lymphoblastic lymphoma/leukemia, and post-transplant lymphoproliferative disease(PTLD) .
* Previously received other BCL-2 protein family inhibitors.
* CLL subject has undergone an allogeneic or autologous stem cell transplant or NHL subject has undergone an allogeneic stem cell transplant.
* Subjects who have received the following treatments within 4 weeks or 5 half-lives before the first dose of LP-108:

  * Antitumor therapies including myelosuppressive chemotherapy, targeted therapy, biological therapy and / or immunotherapy;
  * Any investigational treatment;
  * Patients who have undergone major surgery, severe trauma or radiotherapy.
* Subjects who have received the following treatments within 2 weeks before the first dose of LP-108:

  * Steroids or traditional herbal medicine for antitumor purposes;
  * Strong and moderate CYP3A4/5 inhibitors and inducers, P-gp inhibitors and CYP2C8 sensitive substrates;
  * All drugs that may cause QTc interval prolongation or torsional tachycardia.
* Have had malignancies other than the indications targeted in this study in the past three years, except for basal cell carcinoma of the skin and cervical carcinoma in situ treated radically.
* Any serious and / or uncontrolled systemic disease.
* Poor cardiovascular function, in line with New York Heart Association (NYHA) cardiac function classification ≥ 2 or QTcF greater than 480ms on ≥ 3 independent ECG.
* Disease states where clinical manifestations may be difficult to control, including

  * HIV, HBV, HCV, syphilis positive or active bacterial and fungal infections;
  * Disease affects the central nervous system with obvious symptoms;
  * Autoimmune hemolytic anemia or Idiopathic thrombocytopenic purpura.
* Any gastrointestinal conditions that may severely affect the study drug absorption or pharmacokinetic parameters.
* Patients who were unable to discontinue taking CYP2C8 substrate repaglinide to control type 2 diabetes during the study.
* Subjects who cannot tolerate urine collection, venipuncture, lymph node biopsy, and bone marrow aspiration.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 74 (Estimated)
Dates: Start 2020-05-01 (Actual); Primary Completion 2023-12-01 (Estimated); Study Completion 2023-12-01 (Estimated)

PRIMARY OUTCOMES:
Determination of dose limiting toxicity (DLT), maximum tolerated dose (MTD), recommended phase two dose (RP2D), and lead-in period regimen | Lead-in period (0-4 weeks) plus 3 weeks of study drug administration at the designated cohort dose.
  Protocol-defined events, which can not be attributed by the investigator to a clearly identifiable cause such as tumor progression, underlying illness, concurrent illness, or concomitant medication, will be considered a DLT. Dose limiting toxicities of tumor lysis syndrome observed during the lead-in period will be attributed to the lead-in period.
Number of subjects with adverse events and its frequency | From first dose of study drug administration until 30 days after study drug discontinue.
  Safety Proflie
Determination of plasma peak concentration (Cmax) of LP-108 | Up to Week 37 for LP-108.
  Blood and urine samples for pharmacokinetic analysis of LP-108 will be collected at designated time points.
Determination of Area Under the Curve (AUC) of LP-108 | Up to Week 37 for LP-108.
  Blood and urine samples for pharmacokinetic analysis of LP-108 will be collected at designated time points.
Food Effect - Cmax | Pharmacokinetic (PK) parameter Cmax (maximum plasma concentration of LP-108) between each diet (LP-108 under fasting versus fed conditions)，up to week 8 for LP-108.
  Blood samples for food effect pharmacokinetic analysis of LP-108 will be collected at designated time points
Food Effect - AUC | Pharmacokinetic (PK) parameter AUC (area under the curve of LP-108) between each diet (LP-108 under fasting versus fed conditions)，up to week 8 for LP-108.
  Blood samples for food effect pharmacokinetic analysis of LP-108 will be collected at designated time points

SECONDARY OUTCOMES:
Preliminary efficacy assessment | Designated dose starting week for clinical disease progression and tumor response; and every 4-12 weeks thereafter until the date of first documented progression or date of death from any cause, whichever came first,.assessed up to 24 months.
  Tumor response or clinical disease progression
Minimal residual disease (MRD) | At least 2 months after the CR, CRi criteria for tumor response are first met. Measured up to 24 months after the last subject has enrolled in the study.
  MRD assessed in the peripheral blood and/or bone marrow (BM) either by four color flow cytometry or NGS, will be measured in CLL subjects achieving CR/CRi.

CONTACTS AND LOCATIONS:
Locations (1):
- the First Affiliated Hospital of Nanjing Medical University, Nanjing, Jiangsu, China